CLINICAL TRIAL: NCT03041831
Title: Mobile Health Obesity Wellness Intervention in Rural Older Adults (MOWI): Qualitative Assessment
Brief Title: MOWI Qualitative Assessment
Status: Completed | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, John A. Batsis, MD, Associate Professor of Medicine and of The Dartmouth Institute Geisel School of Medicine at Dartmouth, Dartmouth-Hitchcock Medical Center
Other Study IDs: D16182_1a; K23AG051681 (NIH)
Record Dates: First submitted 2016-11-30; First posted 2017-02-03 (Estimated); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Obesity
Keywords: frail elderly; telemedicine; obesity; rural health; health promotion
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Older adult individual interviews: The investigators will conduct 8 semi-structured 60-minute interviews with patient participants.The goal of these interviews is to determine the acceptability, utility, and perceived value of mobile health (mHealth) in helping older adults overcome barriers to health behavior change.
- Clinician individual interviews: The investigators will conduct 6 semi-structured 60-minute interviews with primary care clinicians who care for older adult populations.The goal of these interviews is to determine the acceptability, utility, and perceived value of mobile health (mHealth) in helping older adults overcome barriers to health behavior change.
- Community leader individual interviews: The investigators will conduct 4 semi-structured 60-minute interviews with community leaders.The goal of these interviews is to determine the acceptability, utility, and perceived value of mobile health (mHealth) in helping older adults overcome barriers to health behavior change.
- Focus group discussions: The investigators will lead four 90-minute focus group discussions consisting of 6-8 older adult participants each. The goal of these focus groups is to determine the acceptability, utility, and perceived value of mobile health (mHealth) in helping older adults overcome barriers to health behavior change.

SUMMARY:
This qualitative study seeks to assess whether mobile health technologies are helpful for older adults. It is the first in a series of four studies whose overarching goal is to conduct a program of pilot research aimed at developing and evaluating a technology-assisted wellness intervention for older adults with obesity who may or may not live in a rural area.

DETAILED DESCRIPTION:
This study is designed and conducted as a series of eighteen individual semi-structured interviews and four focus group discussions. There are three participant groups: 1) older adults (age ≥ 65 years) with diagnosed obesity, 2) primary care clinicians who care for older adults, and 3) community leaders. Focus group discussions are conducted with the older adult cohort only.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65 years;
* Body Mass Index (BMI) ≥ 30kg/m^2;
* Waist circumference ≥88cm in females or ≥102cm in males

Exclusion Criteria:

* Severe mental or life-threatening illness
* Dementia
* Substance use
* History of bariatric surgery
* Suicidal ideation
* Unable to perform measures
* Reside in a nursing home

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Older adult participants screened and recruited primarily in local primary care setting (Department of Community and Family Medicine at Dartmouth Hitchcock Medical Center), as well as through other marketing channels such as posters and radio advertising. Community leaders and clinicians recruited by invitation from the principal investigator.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-08-15 (Actual); Primary Completion 2017-04-28 (Actual); Study Completion 2020-04-28 (Actual)

PRIMARY OUTCOMES:
Technology use in older adults | Up to one year from interview or focus group
  The investigators will record and transcribe each interview and focus group discussion for post-hoc evaluation. The investigators will then use the transcripts to identify themes on perceptions and experience with technology use in older adults.

SECONDARY OUTCOMES:
Determinants of obesity in older adults | Up to one year from interview or focus group
  The investigators will record and transcribe each interview and focus group discussion for post-hoc evaluation. The investigators will then use the transcripts to identify themes related to the secondary outcome. Themes may include (but are not limited to) barriers and facilitators experienced by older adults when they want to lose weight or eat healthier, barriers and facilitators to joining wellness programs, and general availability of options and support.

CONTACTS AND LOCATIONS:
Overall Officials: John A Batsis, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center / Dartmouth Medical School
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Batsis JA, Dokko R, Naslund JA, Zagaria AB, Kotz D, Bartels SJ, Carpenter-Song E. Opportunities to Improve a Mobile Obesity Wellness Intervention for Rural Older Adults with Obesity. J Community Health. 2020 Feb;45(1):194-200. doi: 10.1007/s10900-019-00720-y. PMID 31486958
- [Result] Batsis JA, Zagaria AB, Halter RJ, Boateng GG, Proctor P, Bartels SJ, Kotz D. Use of Amulet in behavioral change for geriatric obesity management. Digit Health. 2019 Jun 21;5:2055207619858564. doi: 10.1177/2055207619858564. eCollection 2019 Jan-Dec. PMID 31258927
- [Result] Batsis JA, Zagaria A, Kotz DF, Bartels SJ, Boateng GG, Proctor PO, Halter RJ, Carpenter-Song EA. Usability Evaluation for the Amulet Wearable Device in Rural Older Adults with Obesity. Gerontechnology. 2018 Sep;17(3):151-159. doi: 10.4017/gt.2018.17.3.003.00. PMID 30631251
- [Result] Batsis JA, Naslund JA, Zagaria AB, Kotz D, Dokko R, Bartels SJ, Carpenter-Song E. Technology for Behavioral Change in Rural Older Adults with Obesity. J Nutr Gerontol Geriatr. 2019 Apr-Jun;38(2):130-148. doi: 10.1080/21551197.2019.1600097. Epub 2019 Apr 11. PMID 30971189
- See also: Mobile Health Obesity Wellness Intervention in Rural Older Adults: Amulet Technology Development & Validation — https://clinicaltrials.gov/ct2/show/NCT03085589?term=NCT03085589&rank=1
- See also: Mobile Health Obesity Wellness Intervention in Rural Older Adults (MOWI): Research Pilot — https://clinicaltrials.gov/show/NCT03104192
- See also: Mobile Health Obesity Wellness Intervention in Rural Older Adults (MOWI): Home-Based Pilot — https://clinicaltrials.gov/show/NCT03104205

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-07-03): https://cdn.clinicaltrials.gov/large-docs/31/NCT03041831/Prot_SAP_ICF_000.pdf